CLINICAL TRIAL: NCT00924027
Title: A Pilot Study of High Dose Rate Brachytherapy in The Radiation Oncology Branch
Brief Title: A Study of Patients Receiving High-Dose Rate Brachytherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Deborah Citrin, M.D., Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090100; 09-C-0100
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2024-09-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cervical Cancer; Endometrial Cancer; Esophageal Cancer; Prostate Cancer; Biliary Cancer
Keywords: Radiation; Cancer; HDR; Brachytherapy; Training
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms; Prostatic Neoplasms; Biliary Tract Neoplasms; Neoplasms | interventions — Radiation; Brachytherapy; Magnetic Resonance Imaging; Tomography, X-Ray Computed; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 1/Radiation Therapy (Experimental): Radiation therapy given as high dose radiation (HDR) Brachytherapy.
  Interventions: Radiation: High Dose Radiation (HDR) Brachytherapy; Diagnostic Test: MRI; Diagnostic Test: CT; Diagnostic Test: PET Scan

INTERVENTIONS:
Radiation: High Dose Radiation (HDR) Brachytherapy — Brachytherapy, the placement of a radioactive source close to a tumor, is a well-established part of the treatment of many malignancies, both for palliative and definitive applications. High dose brachytherapy is useful in many malignancies in order to deliver a high dose of radiation therapy to tumor in a conformal fashion with a rapid dose fall-off with the objective of sparing normal surrounding tissue.
  Other Names: HDR Brachytherapy
Diagnostic Test: MRI — When deemed necessary.
  Other Names: Magnetic Resonance Imaging
Diagnostic Test: CT — Obtained based on the sites of target, as clinical situation dictates and at each follow-up to determine local control.
  Other Names: Computed Tomography
Diagnostic Test: PET Scan — When deemed necessary.
  Other Names: Positron Emission Tomography

SUMMARY:
Background:

* One standard way of giving radiation is to combine external beam treatments with internal brachytherapy treatments, which involve short-range radiation therapy that gives a high dose of radiation directly to a cancer or to the area where cancer cells were removed.
* Brachytherapy is done by placing hollow implant device(s) into the area to be treated and then moving a radiation source into each. The type of device depends on the type of cancer and the site to be treated. These devices can range from hollow applicators and needles to balloon-like equipment.

Objectives:

* To evaluate the quality of the brachytherapy procedure at the National Institutes of Health Radiation Oncology Branch.

Eligibility:

* Patients with cancer who could potentially benefit from high-dose brachytherapy as part of their treatment.

Design:

* In conjunction with their existing treatment, patients will be treated with high-dose brachytherapy as determined appropriate for their particular type of cancer and cancer history.
* Each treatment will take place in the Radiation Oncology Clinic.
* If the patient does not have implant devices, the clinic staff will insert them and check their placement through a computed tomography (CT) scan.
* The calculations to determine the appropriate brachytherapy dose will take a few hours; the brachytherapy treatment itself will take between 10 and 30 minutes.
* The number of brachytherapy treatments will vary according to the individual needs and requirements of each type of cancer and each patient.
* Patients will return to the Radiation Oncology Clinic for follow-up visits at 1, 3, 6, 9, and 12 months after the completion of radiation therapy. Follow-up evaluations will include a medical history and physical examination, assessment of any side effects of radiation therapy, and a repeat of any imaging (i.e., CT, magnetic resonance imaging (MRI), X-ray) that was done at baseline to evaluate the tumor response.

DETAILED DESCRIPTION:
BACKGROUND:

* High dose rate brachytherapy (HDR) is a challenging technique utilized in many malignancies in order to deliver a high dose of radiation therapy to a tumor in a conformal fashion with a rapid dose fall-off with the objective of sparing normal surrounding tissue
* HDR therapy has been targeted to particular subsites as an integral part of either definitive management or palliation for malignancy-related symptoms.

OBJECTIVES:

* The primary objective is to determine the quality of high dose rate brachytherapy implants performed in the radiation oncology branch. An implant will be adequate if 90% of the GTV receives 90% of the dose prescribed and 80% of the Gross Tumor Volume (GTV) receives 85% of the prescribed dose. An implant will be inadequate if the above dose limitations are not met.
* To evaluate local control and late toxicity rates following brachytherapy at the NCI ROB
* To increase the flow of oncology participants requiring brachytherapy to the National Cancer Institute (NCI) Radiation Oncology Branch (ROB), as these participants lend themselves to special study and have unique educational value for the purpose of educating nurses, medical students, residents, physicists, clinical fellows, and physicians.

ELIGIBILITY:

-Participants with cancer who could potentially benefit from the use of high dose rate brachytherapy as a component of their treatment.

DESIGN:

* Participants will undergo appropriate work-up and clinical evaluation to determine if high-dose brachytherapy would be beneficial in either primary treatment or palliation of their disease. Participants will be treated with high-dose brachytherapy appropriately sequenced with other modalities in their treatment regimen. This treatment will be administered in accordance with standard radiation oncology practice and per the ABS (American Brachytherapy Society) guidelines.
* The participants disease status and toxicity outcomes will be documented for a 12-month period at 3-months intervals.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Pathologically confirmed malignancy for which high-dose rate brachytherapy is appropriate as a component of their therapeutic regimen.
  2. Age greater than 18 years of age.
  3. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
  4. Participant must have a primary medical or surgical oncologist in the community or at National Cancer Institute (NCI) who is willing to collaborate with the Radiation Oncology Branch (ROB) staff in the clinical management of the participant.
  5. Participants of childbearing or child- fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated on this study.
  6. Site-specific inclusion criteria (any one or more of the following):

Gynecologic Cancers:

Endometrial cancer

* Participants at a higher risk of recurrence (because of either grade, myometrial invasion, lymphatic vascular space invasion, tumor size, lymph node status, tumor extension, presence or absence of surgical staging)
* Participants who have suffered a recurrence at the vaginal cuff
* Participants who are unable to undergo surgery and must have treatment for an inoperable primary endometrial cancer.

Cervical cancer

* Participants who are unable to undergo surgery and must have treatment for an inoperable primary cervical cancer.
* Participants with locally advanced cervical cancer in whom brachytherapy will be integrated as a boost to external beam radiation either in a palliative or curative setting (definitive or post-operative setting).

Lung cancer

* Participants with an endobronchial component causing symptoms
* Participants who cannot undergo resection because of poor lung function or distant lung metastasis

Breast cancer

* Infiltrating ductal carcinoma or ductal carcinoma in-situ (DCIS), stage T0, T1, and T2 less than or equal to 3.0 cm, N0 and M0,
* Participants benefiting from high dose radiation (HDR) as either as a boost or accelerated partial breast irradiation regimen.

Prostate Cancer

-Participants with localized prostate cancer (T1b-T3b) in whom brachytherapy will be integrated as a boost to external beam radiation or used as monotherapy for definitive management.

EXCLUSION CRITERIA:

1. Cognitively impaired participants who cannot give informed consent.
2. Participants currently receiving concurrent investigational chemotherapeutic agents.
3. Participants receiving concomitant chemotherapy administration in the 5 days preceding brachytherapy (except for gynecological cancer patients who may have received concurrent chemotherapy as a component of their treatment regimen)
4. Pregnant or breast-feeding females are excluded because of the potential mutagenic effects on a developing fetus or newborn.
5. Clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), which in the judgment of the Principal or Associate Investigator would compromise the participant s ability to tolerate this therapy or are likely to interfere with the study procedures or results.
6. Participants who are in the estimation of the PI, deemed unable or unlikely to adhere to protocol treatment.
7. Abnormal bleeding times or active anti-coagulation therapy.

   * platelets less than 100,000 per mm(3)
   * Prothrombin time (PT)/Partial thromboplastin time (PTT) greater than 1.5 the upper normal limit (UNL)
8. Any participant or tumor/anatomical factors that may prevent brachytherapy apparatus from being properly and safely inserted and positioned and from radiation therapy being administered per American Brachytherapy Society (ABS) guidelines.
9. Participants whose malignancy has one or more of the following site-specific criteria disqualifying them from the study:

1. Breast cancer:

* Participants inappropriate for standard breast conservation therapy (Multicentric disease, inability to achieve clear margins);
* male participants with breast cancer
* autoimmune disorders, including systemic lupus erythematosus (SLE), Scleroderma, etc.
* distant metastases;

  2. Prostate cancer:
* distant metastases
* lymph node metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-04-14 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2025-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Citrin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Creutzberg CL, van Putten WL, Koper PC, Lybeert ML, Jobsen JJ, Warlam-Rodenhuis CC, De Winter KA, Lutgens LC, van den Bergh AC, van de Steen-Banasik E, Beerman H, van Lent M. Surgery and postoperative radiotherapy versus surgery alone for patients with stage-1 endometrial carcinoma: multicentre randomised trial. PORTEC Study Group. Post Operative Radiation Therapy in Endometrial Carcinoma. Lancet. 2000 Apr 22;355(9213):1404-11. doi: 10.1016/s0140-6736(00)02139-5. PMID 10791524
- [Background] Kocak Z, Ozkan H, Adli M, Garipagaoglu M, Kurtman C, Cakmak A. Intraluminal brachytherapy with metallic stenting in the palliative treatment of malignant obstruction of the bile duct. Radiat Med. 2005 May;23(3):200-7. PMID 15940068
- [Background] Perez CA, Grigsby PW, Castro-Vita H, Lockett MA. Carcinoma of the uterine cervix. I. Impact of prolongation of overall treatment time and timing of brachytherapy on outcome of radiation therapy. Int J Radiat Oncol Biol Phys. 1995 Jul 30;32(5):1275-88. doi: 10.1016/0360-3016(95)00220-S. PMID 7635767
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0100.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Gynecologic (Endometrial & Cervical): Participants received brachytherapy to the vaginal cuff or to the cervical or uterine tumor. Brachytherapy, the placement of a radioactive source close to a tumor, is a well-established part of the treatment of many malignancies, both for palliative and definitive applications. Participants will be treated with high-dose brachytherapy according to standard oncology practice and the American Brachytherapy Society (ABS) guidelines. Treatment will vary depending on the site of disease treated.
- Pulmonary; Breast: No participants were accrued to this group.
- Prostate: Participants received brachytherapy to the prostate.
Period: Overall Study
Arm/Group | Gynecologic (Endometrial & Cervical) | Pulmonary | Breast | Prostate
Started | 28 | 0 | 0 | 15
Started Brachytherapy | 27 | 0 | 0 | 14
Completed Brachytherapy | 26 | 0 | 0 | 14
Follow-up Period Active | 0 | 0 | 0 | 0
Follow-Up Period Completed | 20 | 0 | 0 | 14
Completed | 20 | 0 | 0 | 14
Not Completed | 8 | 0 | 0 | 1
Not completed — Lost to Further Follow-Up | 4 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1
Not completed — Withdrawal: Refused further treatment | 1 | 0 | 0 | 0
Not completed — Withdrawal: Refused to start treatment | 1 | 0 | 0 | 0
Not completed — Withdrawal: Refused further follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were accrued to the Pulmonary and Breast Group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gynecologic (Endometrial & Cervical) | Pulmonary | Breast | Prostate | Total
Number analyzed (Participants) | 28 | 0 | 0 | 15 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0 | 0
  Between 18 and 65 years | 14 |  |  | 4 | 18
  >=65 years | 14 |  |  | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (12.4) |  |  | 68.4 (7.1) | 66.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 |  |  | 0 | 28
  Male | 0 |  |  | 15 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  |  | 0 | 1
  Not Hispanic or Latino | 27 |  |  | 15 | 42
  Unknown or Not Reported | 0 |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 |  |  | 0 | 1
  Asian | 4 |  |  | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0 | 0
  Black or African American | 4 |  |  | 6 | 10
  White | 19 |  |  | 8 | 27
  More than one race | 0 |  |  | 0 | 0
  Unknown or Not Reported | 0 |  |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 |  |  | 15 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Adequate High-Quality Brachytherapy Implants Reported Per Strata (Four Body Sites) and Combined Overall
Description: An implant is adequate if 90% of the Gross Tumor Volume (GTV) receives 90% of the dose prescribed and 80% of the Clinical Tumor Volume (CTV) receives 85% of the prescribed dose. An implant is inadequate if the above criteria is not met. A GTV only applies to certain disease sites such as gynecologic cancer that have not been removed by surgery and CTV applies to prostate or gynecologic cancer that have been removed surgically.
Time Frame: All participants were assessed 1 week after last dose of high dose radiation (HDR) brachytherapy, an average of 1 week (no range).
Population: As pre-specified by the protocol, this outcome measure is reported per strata (body sites). No participants were accrued to the pulmonary and breast body sites. 27/28 participants were analyzed in the gynecologic group and 14/15 participants were analyzed in the prostate group because one participant in each group withdrew and refused to start treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Gynecologic (Endometrial & Cervical), and Prostate combined. No participants were accrued to the pulmonary and breast group. All participants who received HDR brachytherapy were assessed 1-week after last dose.
Arm/Group | Gynecologic (Endometrial & Cervical) | Pulmonary | Breast | Prostate | Overall
Number analyzed (Participants) | 27 | 0 | 0 | 14 | 41
Participants | 27 | 0 | 0 | 14 | 41

2. Secondary Outcome: Number of Prostate Participants With Local Control
Description: Local control of the prostate is defined as Biochemical recurrence. Biochemical recurrence is a serum prostatic specific antigen (PSA) more than 2 ng/dL above the post brachytherapy nadir, measured by at least 2 PSA measurements separated by 1 month, and the National Comprehensive Cancer Network (NCCN) guidelines.
Time Frame: Assessed at 12 months after radiation
Population: As pre-specified by the protocol, this outcome measure is reported per strata (body sites). No participants were accrued to the pulmonary and breast body sites. 14/15 participants were analyzed in the prostate group because one participant withdrew and refused to start treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Prostate
Number analyzed (Participants) | 14
Participants
  Biochemical recurrence | 0
  No recurrence | 14
  Not evaluable | 0

3. Secondary Outcome: Number of Participants With Local Control Reported Per Strata (Body Sites) and Combined Overall
Description: Local control is defined as Complete Response (CR), Partial Response (PR) or Stable Disease (SD) of the treated site. In diseases where targets can be imaged, response will be measured using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria only for local sites. Complete Response is disappearance of the target lesion. Partial Response is at least a 30% decrease in the sum of the longest diameter (LD) of the target lesion taking into account the baseline sum LD. Stable Disease does not qualify for CR, PR, or progression. Progression is interval increase in the maximal dimension of the target lesion. Scoring of local control at each treated site will be based on Response Evaluation Criteria in Solid Tumor (RECIST) criteria. Each site will be scored separately (Only for local sites) and the number of participants with CR, PR, SD will be determined.
Time Frame: Assessed at 12 months after radiation
Population: As pre-specified by the protocol, this outcome measure is reported per strata (body sites). The prostate group were intentionally reported separately because the assessment for local control is different between the prostate (e.g., biochemical recurrence) group and gynecologic (e.g., imaging) group. No participants were accrued to the pulmonary and breast body sites. 27/28 participants were analyzed in the gynecologic group because one participant withdrew and refused to start treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Gynecologic (Endometrial & Cervical) | Pulmonary | Breast | Overall
Number analyzed (Participants) | 27 | 0 | 0 | 27
Participants
  Complete Response | 25 | 0 | 0 | 25
  Partial Response | 0 | 0 | 0 | 0
  Stable Disease | 0 | 0 | 0 | 0
  Not Evaluable | 2 | 0 | 0 | 2

4. Secondary Outcome: Number of Grades 0-5 Late Toxicity Reported Per Strata (Body Sites) and Combined Overall
Description: The Radiation Therapy Oncology Group (RTOG)/European Organization for Research and Treatment of Cancer (EORTC) Radiation Morbidity Scoring Scheme was used to score late toxicity following brachytherapy. Late toxicities are graded 0-5. Grade 0 is no symptoms. Grade 1 is mild/slight symptoms. Grade 2 is moderate. Grade 3 is severe. Grade 4 is severe/life-threatening. And Grade 5 is toxicity related to death.
Time Frame: Date treatment consent signed to date off study, approximately 159 months and 21 days.
Population: as for outcome 1
Measure: Number; unit: Toxicities
Arm/Group | Gynecologic (Endometrial & Cervical) | Pulmonary | Breast | Prostate | Overall
Number analyzed (Participants) | 27 | 0 | 0 | 14 | 41
Toxicities
  Grade 0 | 0 |  |  | 0 | 0
  Grade 1 | 8 |  |  | 17 | 25
  Grade 2 | 14 |  |  | 15 | 29
  Grade 3 | 1 |  |  | 1 | 2
  Grade 4 | 1 |  |  | 0 | 1
  Grade 5 | 0 |  |  | 0 | 0

5. Secondary Outcome: Number of Participants Accrued Who Received Brachytherapy Each Year
Description: To help understand and increase the flow of participants receiving brachytherapy, the number of participants who received brachytherapy each year are reported.
Time Frame: Approximately 16 years
Population: No participants were accrued to the pulmonary and breast group. 27/28 participants were analyzed in the gynecologic group and 14/15 participants were analyzed in the prostate group because one participant in each group withdrew and refused to start treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Gynecologic (Endometrial & Cervical) | Pulmonary | Breast | Prostate | Overall
Number analyzed (Participants) | 27 | 0 | 0 | 14 | 41
Participants
  Year 2009 | 3 |  |  | 0 | 3
  Year 2010 | 2 |  |  | 0 | 2
  Year 2011 | 2 |  |  | 0 | 2
  Year 2012 | 12 |  |  | 0 | 12
  Year 2013 | 4 |  |  | 0 | 4
  Year 2014 | 2 |  |  | 0 | 2
  Year 2015 | 1 |  |  | 0 | 1
  Year 2016 | 1 |  |  | 3 | 4
  Year 2017 | 0 |  |  | 1 | 1
  Year 2018 | 0 |  |  | 7 | 7
  Year 2019 | 0 |  |  | 1 | 1
  Year 2020 | 0 |  |  | 0 | 0
  Year 2021 | 0 |  |  | 1 | 1
  Year 2022 | 0 |  |  | 0 | 0
  Year 2023 | 0 |  |  | 0 | 0
  Year 2024 | 0 |  |  | 1 | 1

6. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria (CTC) v3.0
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria (CTC v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Assessed at 12 months after radiation
Population: No participants were accrued to the pulmonary and breast group. And no participants were assessed for adverse events in the prostate group using the CTCv3.0. 26/28 participants were analyzed in the gynecologic group because one participant withdrew and refused to start treatment, and one participant did not complete brachytherapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Gynecologic (Endometrial & Cervical) | Pulmonary | Breast | Prostate | Overall
Number analyzed (Participants) | 25 | 0 | 0 | 0 | 25
Participants | 22 | 0 | 0 | 0 | 22

7. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Radiation Therapy Oncology Group (RTOG)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the RTOG. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Assessed at 12 months after radiation
Population: No participants were accrued to the pulmonary and breast group. 27/28 participants were analyzed in the gynecologic group and 4/15 participants were analyzed in the prostate group because one participant refused to start treatment in each group.
Measure: Count of Participants; unit: Participants
Arm/Group | Gynecologic (Endometrial & Cervical) | Pulmonary | Breast | Prostate | Overall
Number analyzed (Participants) | 27 | 0 | 0 | 14 | 41
Participants | 19 | 0 | 0 | 11 | 30

ADVERSE EVENTS:
Time Frame: Start date of brachytherapy to date off study, an average of 13 months.
Description: Adverse events (AE) were graded by the *CTCv3.0 from the start date of brachytherapy through 30 days after the intervention was last administered and ~RTOG from 30 days after the intervention was last administered to off study, as noted.
  27/28 participants were analyzed in the gynecologic group and 14/15 participants were analyzed in the prostate group because one participant refused to start treatment in each group.
Arm/Group | Gynecologic (Endometrial & Cervical) | Pulmonary | Breast | Prostate
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/0 | 0/0 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/0 | 0/0 | 0/14
Other Adverse Events (participants affected / at risk) | 22/27 | 0/0 | 0/0 | 11/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gynecologic (Endometrial & Cervical) (N=27) | Pulmonary (N=0) | Breast (N=0) | Prostate (N=14)
*Anorexia (Metabolism and nutrition disorders) | 1 (1) | NA | NA | 0 (0)
*Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 (7) | NA | NA | 0 (0)
*Constipation (Gastrointestinal disorders) | 1 (1) | NA | NA | 0 (0)
*Diarrhea (Gastrointestinal disorders) | 8 (8) | NA | NA | 0 (0)
*Fatigue (asthenia, lethargy, malaise) (General disorders) | 7 (7) | NA | NA | 0 (0)
*Nausea (Gastrointestinal disorders) | 5 (6) | NA | NA | 0 (0)
*Infection with normal ANC or Grade 1 or 2 neutrophils: Urinary tract NOS (Infections and infestations) | 5 (7) | NA | NA | 0 (0)
*Pain - Other (Specify, right and left groin) (Reproductive system and breast disorders) | 1 (1) | NA | NA | 0 (0)
*Intra-operative injury:: Vulva (Injury, poisoning and procedural complications) | 1 (1) | NA | NA | 0 (0)
*Pain:: Abdomen NOS (Gastrointestinal disorders) | 4 (4) | NA | NA | 0 (0)
*Pain:: Back (Musculoskeletal and connective tissue disorders) | 2 (2) | NA | NA | 0 (0)
*Pain:: Head/Headache (Nervous system disorders) | 1 (1) | NA | NA | 0 (0)
*Pain:: Muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | NA | 0 (0)
*Pain:: Pain NOS (General disorders) | 1 (1) | NA | NA | 0 (0)
*Pain:: Pelvis (Reproductive system and breast disorders) | 2 (2) | NA | NA | 0 (0)
*Pain:: Perineum (Gastrointestinal disorders) | 1 (1) | NA | NA | 0 (0)
*Pain:: Urethra (Renal and urinary disorders) | 1 (2) | NA | NA | 2 (2)
*Pain:: Vagina (Reproductive system and breast disorders) | 6 (6) | NA | NA | 0 (0)
*Platelets (Blood and lymphatic system disorders) | 1 (1) | NA | NA | 0 (0)
*Potassium, serum low (hypokalemia) (Metabolism and nutrition disorders) | 1 (2) | NA | NA | 0 (0)
*Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (3) | NA | NA | 0 (0)
*Urinary frequency/urgency (Renal and urinary disorders) | 3 (4) | NA | NA | 0 (0)
*Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1) | NA | NA | 0 (0)
*Urine color change (Renal and urinary disorders) | 3 (3) | NA | NA | 0 (0)
*Dizziness (Nervous system disorders) | 1 (1) | NA | NA | 0 (0)
*Neuropathy:: sensory (Nervous system disorders) | 1 (2) | NA | NA | 0 (0)
*Vaginal discharge (non-infectious) (Reproductive system and breast disorders) | 3 (3) | NA | NA | 0 (0)
*Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | NA | NA | 0 (0)
*Vaginitis (not due to infection) (Reproductive system and breast disorders) | 2 (2) | NA | NA | 0 (0)
*Vomiting (Gastrointestinal disorders) | 3 (3) | NA | NA | 0 (0)
*Incontinence, urinary (Renal and urinary disorders) | 1 (1) | NA | NA | 0 (0)
*Hemorrhage, GU:: Vagina (Reproductive system and breast disorders) | 8 (11) | NA | NA | 0 (0)
*Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | NA | NA | 0 (0)
*Cystitis (Renal and urinary disorders) | 2 (2) | NA | NA | 0 (0)
*Dehydration (Metabolism and nutrition disorders) | 1 (1) | NA | NA | 0 (0)
*Hemoglobin (Blood and lymphatic system disorders) | 4 (4) | NA | NA | 0 (0)
*Hemorrhoids (Gastrointestinal disorders) | 1 (1) | NA | NA | 0 (0)
*Incontinence, anal (Gastrointestinal disorders) | 1 (1) | NA | NA | 0 (0)
*Hypertension (Vascular disorders) | 4 (6) | NA | NA | 0 (0)
Lower gastrointestinal tract (Gastrointestinal disorders) | 5 (5) | NA | NA | 7 (7)
Leukocytes or white blood cells (Blood and lymphatic system disorders) | 1 (1) | NA | NA | 1 (1)
Genitourinary (Renal and urinary disorders) | 8 (8) | NA | NA | 9 (10)
Bladder (Renal and urinary disorders) | 8 (8) | NA | NA | 8 (10)
Small and large intestine (Gastrointestinal disorders) | 5 (6) | NA | NA | 3 (5)
Mucous Membrane (Skin and subcutaneous tissue disorders) | 9 (14) | NA | NA | 0 (0)
Skin (Skin and subcutaneous tissue disorders) | 5 (7) | NA | NA | 0 (0)
Subcutaneous Tissue (Skin and subcutaneous tissue disorders) | 10 (15) | NA | NA | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT00924027/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT00924027/ICF_001.pdf